CLINICAL TRIAL: NCT00323388
Title: Identification of Risk Allels for Prostate Cancer
Status: Withdrawn | Type: Observational
Why Stopped: No subjects enrolled and this is not a clinical trial. Was inadvertently entered in the system.
Sponsor: University of New Mexico (Other)
Responsible Party: John Scariano; Principal Investigator, Universtiy of New Mexico
Other Study IDs: HRRC 04-458
Record Dates: First submitted 2006-05-05; First posted 2006-05-09 (Estimated); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Identification of Risk Allels for Prostate Cancer

DETAILED DESCRIPTION:
As above.

ELIGIBILITY:
Inclusion Criteria:

* Patients with prostate cancer.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-11 (Actual); Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Scariano, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States